CLINICAL TRIAL: NCT06657170
Title: Hidden Slow Conduction Ablation for Recurrent Atrial Fibrillation: Unmasking the Arrhythmogenic Substrate
Brief Title: Hidden Slow Conduction Ablation for Recurrent Atrial Fibrillation: Unmasking the Arrhythmogenic Substrate (Unmask-AF)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Medico Teknon (Other)
Responsible Party: Principal Investigator, Antonio Berruezo, MD, PhD, Director of Electrophysiology unit, Centro Medico Teknon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unmask-AF
Record Dates: First submitted 2024-08-22; First posted 2024-10-24 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Atrial Fibrillation
Keywords: Catheter Ablation; Re-do Procedures; Hidden Slow Conduction; Functional Substrate Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: This is a two-arm, single-center, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PV reconnection + HSC ablation (Experimental): Patients undergoning pulmunary veins (PV) reconnection checking and ablation plus identification and ablation of hidden sites of slow conduction (HSC)
  Interventions: Procedure: Pulmunary veins reconnection plus hidden slow conduction ablation
- PV reconnection ablation only (Active Comparator): Patients undergoning PV reconnection checking and ablation only.
  Interventions: Procedure: Pulmunary veins (PV) reconnection ablation only

INTERVENTIONS:
Procedure: Pulmunary veins reconnection plus hidden slow conduction ablation — Ablation of pulmonary veins reconnections plus the search and ablation of hidden slow conductions sites (HSC) in the left atrium.
  HSC sites are defined as EGMs showing highly fragmented or double electrograms in response atrial triple extrastimulus, presenting normal or fractionated electrogram in the sinus rhythm.
  After checking for PV's conduction breakthroughs, point-by point ablation targeting HSC-EGMs will be performed.
  The end point for HSC+ ablation will be reached with loss of local capture at a given lesion, pacing from the ablation catheter at high output (10V·2ms).
  Arms: PV reconnection + HSC ablation
Procedure: Pulmunary veins (PV) reconnection ablation only — Each vein will be re-assessed by observing PV potentials along the PV ostia and by pacing from the distal bipole of the ablation catheter (10mA at 2ms) within the lesion set with failed capture of the left atrium. In case of PVs reconnection touch-up applications will be performed at the earliest potential site, identified by comparing far-field atrial EGM to near-field local EGM timing, until isolation will be achieved (entrance and exit block).
  Arms: PV reconnection ablation only

SUMMARY:
Over recent years, pulmonary vein isolation (PVI) procedures have demonstrated progressively enhanced efficacy and safety, resulting in a substantial increase in the number of atrial fibrillation ablations, not only as a first-line treatment but also for repeat procedures. However, there is still a notable lack of randomized evidence in this area, which limits guidance and decision-making in clinical practice. Recently, the investigators found that employing short-coupled atrial extrastimuli revealed highly fragmented or double atrial evoked electrograms (EGMs) in AF patients, termed as hidden slow conduction (HSC). Identifying HSC sites may provide insight into the early identification of the arrhythmogenic substrate, offering a potential target for ablation This multi-center, prospective, randomized, controlled trial will include two arms: one investigational (PV reconnection + HSC) and one control (PV reconnection). All the subjects will be followed for 12 months after the ablation procedure.

The aim of our study is to investigate the impact of ablating HSC sites on arrhythmia recurrence in repeat ablation procedures. The hypothesis is that the additional ablation of HSC zones may improve the freedom from atrial arrhythmia recurrence after repeat ablation procedure.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent paroxysmal AF (continuous AF episode lasting longer than 30 s but terminating spontaneously or with intervention within 7 days of onset), recurrent persistent AF (continuous AF episode lasting longer than 7 days but < 1 year) and recurrent long standing persistent AF (continuous AF ≥1 year in duration, in patients where rhythm control management is being pursued)
* Previous PVI procedure
* Age > 40 years
* Willing and capable of providing consent
* Able and willing to comply with all follow-up testing and requirements

Exclusion Criteria:

* Additional left atrial ablations during the previous procedures (es. posterior wall isolation, anterior line, roof line, CFAE and others)
* Acute illness, active systemic infection, or sepsis
* Presence of intracardiac thrombus, myxoma, tumor, interatrial baffle or patch or other abnormality that precludes catheter introduction or manipulation.
* Severe mitral regurgitation
* Women who are pregnant, lactating, or who are planning to become pregnant during the course of the clinical investigation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Atrial arrhythmias recurrence | up to 12 moths
  The primary endpoint of the study aims to establish the impact of targeting HSC sites alongside PV gaps in repeat ablation procedures for patients with recurrent AF. Specifically evaluating the freedom from atrial tachyarrhythmia recurrence (documented AF/AT/AFL lasting at least 30s).

SECONDARY OUTCOMES:
Burden of atrial arrhythmias | up to 12 moths
  Arrhythmic burden (average percentage of time in AF/AT in 24h Holter)
incidence of periprocedural complications (pericardial effusion) | up to 12 months
  incidence of periprocedural complications such as pericardial effusion
Use of antiarrhythmic drugs | up to 12 months
  Use of antiarrhythmic drugs after the blanking period of 60 days.
incidence of periprocedural complications (peripheral complication) | up to 12 moths
  incidence of periprocedural complications such as peripheral complication
incidence of periprocedural complications (transient ischemic attack or stroke) | up to 12 months
  incidence of periprocedural complications such as transient ischemic attack or stroke

OTHER OUTCOMES:
Concentration of intramyocardial fat (inFAT) into the HSC points | up to 12 months
  Concentration of intramyocardial fat (inFAT) into the atrial area where we found the HSC points
Procedure features | up to 12 months
  procedure time
Atrial arrhythmias first recurrence | up to 12 months
  Evaluation of the atrial arrhythmias recurrence in patients with isolated PVs underwent HSC sites ablation
Left atrial wall thickness (LAWT) measurement into the HSC points | up to 12 months
  Left atrial wall thickness (LAWT) measurement into the atrial areas where we found the HSC points
procedure features | up to 12 months
  fluoroscopy time
procedure features | up to 12 months
  fluoroscopy dose
procedure features | up to 12 months
  number of radiofrequency (RF) applications
procedure times | up to 12 months
  radiofrequency (RF) total delivery time

REFERENCES:
- [Result] Pokushalov E, Romanov A, De Melis M, Artyomenko S, Baranova V, Losik D, Bairamova S, Karaskov A, Mittal S, Steinberg JS. Progression of atrial fibrillation after a failed initial ablation procedure in patients with paroxysmal atrial fibrillation: a randomized comparison of drug therapy versus reablation. Circ Arrhythm Electrophysiol. 2013 Aug;6(4):754-60. doi: 10.1161/CIRCEP.113.000495. Epub 2013 Jun 7. PMID 23748210
- [Result] Saglietto A, Falasconi G, Soto-Iglesias D, Francia P, Penela D, Alderete J, Viveros D, Bellido AF, Franco-Ocana P, Zaraket F, Turturiello D, Marti-Almor J, Berruezo A. Assessing left atrial intramyocardial fat infiltration from computerized tomography angiography in patients with atrial fibrillation. Europace. 2023 Dec 6;25(12):euad351. doi: 10.1093/europace/euad351. PMID 38011712
- [Result] Silva Garcia E, Lobo-Torres I, Fernandez-Armenta J, Penela D, Fernandez-Garcia M, Gomez-Lopez A, Soto-Iglesias D, Fernandez-Rivero R, Vazquez-Garcia R, Acosta J, Bisbal F, Cano-Calabria L, Berruezo A. Functional mapping to reveal slow conduction and substrate progression in atrial fibrillation. Europace. 2023 Nov 2;25(11):euad246. doi: 10.1093/europace/euad246. PMID 37961921